CLINICAL TRIAL: NCT00000948
Title: A Randomized, Open Label Phase II Study of Subcutaneous Interleukin-2 (Proleukin) Plus Antiretroviral Therapy vs. Antiretroviral Therapy Alone in Patients With HIV Infection and at Least 350 CD4+ Cells/mm3
Brief Title: Effects of Giving Interleukin-2 (IL-2) Plus Anti-HIV Therapy to HIV-Positive Patients With CD4 Cell Counts of at Least 350 Cells/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRP 021B; 10465 (Registry Identifier: DAIDS ES); THAILAND
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Injections, Subcutaneous; Interleukin-2; Dose-Response Relationship, Drug; Drug Therapy, Combination; CD4 Lymphocyte Count; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — aldesleukin

ARMS (2):
- 1 (Experimental): Participants will be broken into 3 groups. Each group will receive ART and escalating doses of aldesleukin. All participants will then receive that maximum tolerated dose of aldesleukin.
  Interventions: Drug: Aldesleukin; Drug: ART
- 2 (Active Comparator): All participants will receive ART
  Interventions: Drug: ART

INTERVENTIONS:
Drug: Aldesleukin — Il-2
  Arms: 1
Drug: ART — antiretroviral therapy for the treatment of HIV

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of giving IL-2 plus anti-HIV (antiretroviral) therapy to HIV-positive patients with CD4 cell counts (cells of the immune system that fight infection) of at least 350 cells/mm3. This study will also examine the ability of antiretroviral therapy combined with IL-2 to boost the immune system.

IL-2, given through injection under the skin, in combination with anti-HIV therapy can increase CD4 cell counts. This study examines 3 doses of IL-2 in order to determine the safest and most effective dose to use.

DETAILED DESCRIPTION:
Interleukin-2 administered subcutaneously, in combination with antiretrovirals, results in an increased CD4+ cell count that might impact upon HIV disease progression. A Phase III trial involving large numbers of HIV-positive patients is the next step in the development process. To develop appropriate clinical experience with this combination, this Phase II trial will allow administration of IL-2 plus antiretroviral therapy to a small number of patients in sites being considered for the Phase III trial.

Patients receive antiretrovirals alone or antiretrovirals plus IL-2 given subcutaneously. Three doses of IL-2 are studied, with 12 patients evaluated at each dose. When at least 9 of the first 12 patients complete the 5-day dosing period without dose-limiting toxicity, the next 12 patients are treated at the next highest dose every 12 hours for 5 days every 8 weeks; when this dose is tolerated, the last 12 patients randomized receive the highest study dose every 12 hours for 5 days every 8 weeks. Patients enrolled at the first two doses of IL-2 who complete three courses of treatment have their dose escalated to a maximum of the highest study dose.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a CD4 cell count greater than or equal to 300 cells/mm3.
* Have no AIDS-defining illnesses.
* Are at least 18 years old.
* Have been on antiretroviral therapy for at least 7 days prior to study entry.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Abuse alcohol or drugs, or have any serious psychiatric or medical illnesses that would affect their safety or ability to complete the study.
* Have a history of cancer (other than Kaposi's sarcoma), an AIDS-defining illness, a central nervous system abnormality, or an autoimmune/inflammatory disease.
* Are pregnant or breast-feeding.
* Have ever received IL-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 1998-02; Primary Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
CD4 count | Throughout study
Laboratory and clinical adverse events | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungthum, Study Chair
Locations (2):
- Thailand (2):
  - Chulalongkorn Univ. Hosp. C603-010 CRS, Bangkok, Ratchathewi
  - Siriraj Hospital C603-020 CRS, Bangkok, Ratchathewi